CLINICAL TRIAL: NCT03686540
Title: Costs of the Patient's Stay Under ExtraCorporeal Membrane Oxygenation From the Hospital Point of View: a Pilot Study at the Rennes University Hospital Center
Acronym: ECMONOMY
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_3042_ECMONOMY
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: ExtraCorporeal Membrane Oxygenation
MeSH Terms: interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ExtraCorporeal Membrane Oxygenation (ECMO) — The objective of this study is to determine the average cost of stay of a patient supported by ExtraCorporeal Membrane Oxygenation from the point of view of the hospital facility, during the hospitalization in which the ECMO was implanted.

SUMMARY:
The objective of this study is to determine the average cost of stay of a patient supported by ExtraCorporeal Membrane Oxygenation from the point of view of the hospital facility, during the hospitalization in which the ECMO was implanted.

ELIGIBILITY:
Inclusion Criteria:

All patients ≥18 years old who have benefited from an ECMO (no type, no indication) between 2004 and 2016 at the Rennes University Hospital, identified in the database of the Rennes University Hospital Center will be included in this study.

Exclusion Criteria:

Neither

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who benefited from an ECMO at Rennes University Hospital Center
Sampling Method: Non-Probability Sample
Enrollment: 620 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Average net costs | 1 day of inclusion
  Average net costs (total and by expense) for the hospital facility (Rennes University Hospital) of the initial hospitalization. The average net cost for the institution is defined as the average difference between the production costs for the hospital and the incomes donated to the institution by the Health Insurance.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rennes, Rennes, Brittany Region, France